CLINICAL TRIAL: NCT05147818
Title: Risk Factors for Acute Kidney Injury in Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Salah Ali, Principal investigator, Assiut University
Other Study IDs: SSA
Record Dates: First submitted 2021-11-27; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: 200 Diabetic patients of 18 year and older (either type 1or 2) presented by AKI based on KIDIGO Definition & Staging. KDIGO definition of AKI: Increase in serum creatinine by ≥0.3 mg/dL (≥26.5 µmol/L) within 48 h, or Increase in serum creatinine to ≥1.5 times baseline that is known or presumed to have occurred within the prior 7 days, or Urine volume <0.5 mL/kg/h for 6 h.
  KDIGO staging of AKI: (1) stage 1: Serum creatinine 1.5-1.9 × baseline or ≥0.3 mg/dL (≥26.5 µmol/L) increase / Urine output <0.5 mL/kg/h for 6-12 h (2) stage 2; Serum creatinine 2.0-2.9 × baseline / Urine output <0.5 mL/kg/h for ≥12 h (3) stage 3: Serum creatinine 3.0 × baseline, increase in serum creatinine to ≥4.0 mg/dL (≥353.6 µmol/L), initiation of renal replacement therapy, or, in patients <18 years, decrease in eGFR to <35 mL/min per 1.73 m2 / Urine output <0.3 mL/kg/h for ≥24 h or anuria for ≥12 h .
  Interventions: Other: CBC ,renal function tests , fundus Examination
- Controls: 200 Diabetic patients of 18 year and older with no AKI (either type 1or 2) Matched to controls in age ,sex

INTERVENTIONS:
Other: CBC ,renal function tests , fundus Examination — Laboratory investigations
  Other Names: ECG
  Groups: Cases

SUMMARY:
incidence of AKI in diabetic patients seems to be influenced by multiple risk Factors like severe infections, elderly, poor diabetic control, previous AKI, chronic kidney disease and drugs like SGLT2-I increase risk of AKI in diabetic patients.

DETAILED DESCRIPTION:
The incidence and prevalence of diabetes mellitus (DM) have increased over the last 20 years. The defining feature of diabetes mellitus (DM) is the presence of hyperglycaemia . mostly due to the progressively increasing prevalence of obesity and the metabolic syndrome, Current prevalence of DM worldwide is estimated to be about 390 million people . The Cardiovascular complications increase morbidity and mortality in diabetic patients. About 40% of end-stage renal disease on regular dialysis are diabetic . Acute kidney injury (AKI) Is a fundamental problem in hospitalized patients; its incidence has been reaching 20% in middle-Europe . About 50% of patients presented with AKI are found to be diabetic ; which may indicate a direct relationship between the two conditions. In 2012, a clinical practice guideline published by Kidney Disease: Improving Global Outcomes (KDIGO) provided a unifying definition and staging system for AKI . On the other hand, incidence of AKI in diabetic patients seems to be influenced by multiple risk Factors like severe infections, elderly, poor diabetic control, previous AKI, chronic kidney disease and drugs like SGLT2-I increase risk of AKI in diabetic patients. We aim in this study to identify the most common risk factors for AKI in diabetic patients and how those risk factors affect morbidity and mortality in patients with DM who developed AKI.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion criteria for the cases :

200 Diabetic patients of 18 year and older (either type 1or 2) presented by AKI based on KIDIGO Definition & Staging. KDIGO definition of AKI: Increase in serum creatinine by ≥0.3 mg/dL (≥26.5 µmol/L) within 48 h, or Increase in serum creatinine to ≥1.5 times baseline that is known or presumed to have occurred within the prior 7 days, or Urine volume <0.5 mL/kg/h for 6 h.

KDIGO staging of AKI: (1) stage 1: Serum creatinine 1.5-1.9 × baseline or ≥0.3 mg/dL (≥26.5 µmol/L) increase / Urine output <0.5 mL/kg/h for 6-12 h (2) stage 2; Serum creatinine 2.0-2.9 × baseline / Urine output <0.5 mL/kg/h for ≥12 h (3) stage 3: Serum creatinine 3.0 × baseline, increase in serum creatinine to ≥4.0 mg/dL (≥353.6 µmol/L), initiation of renal replacement therapy, or, in patients <18 years, decrease in eGFR to <35 mL/min per 1.73 m2 / Urine output <0.3 mL/kg/h for ≥24 h or anuria for ≥12 h .

Inclusion criteria for matched controls 200 Diabetic patients of 18 year and older with no AKI (either type 1or 2)

Exclusion Criteria:

Exclusion criteria for cases and controls:

1. Non-Diabetic patients with AKI
2. Diabetic patients with:

   * HBS Ag, HCV, HIV
   * Active Lupus
   * Active Malignancy
   * Acute or Chronic Liver Disease
   * Acute poisoning

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients aged from 18 year and older Diabetic patients.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Identify risk factors for Acute kidney injury in diabetic patients | 2 years
  Identify risk factors for Acute kidney injury in d iabetic patients

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. (2) Classification and diagnosis of diabetes. Diabetes Care. 2015 Jan;38 Suppl:S8-S16. doi: 10.2337/dc15-S005. No abstract available. PMID 25537714
- [Background] Aziz Z, Absetz P, Oldroyd J, Pronk NP, Oldenburg B. A systematic review of real-world diabetes prevention programs: learnings from the last 15 years. Implement Sci. 2015 Dec 15;10:172. doi: 10.1186/s13012-015-0354-6. PMID 26670418
- [Background] Mima A. Diabetic nephropathy: protective factors and a new therapeutic paradigm. J Diabetes Complications. 2013 Sep-Oct;27(5):526-30. doi: 10.1016/j.jdiacomp.2013.03.003. Epub 2013 Apr 22. PMID 23619194
- [Background] Bienholz A, Wilde B, Kribben A. From the nephrologist's point of view: diversity of causes and clinical features of acute kidney injury. Clin Kidney J. 2015 Aug;8(4):405-14. doi: 10.1093/ckj/sfv043. Epub 2015 Jul 9. PMID 26251707
- [Background] DeFronzo RA, Reeves WB, Awad AS. Pathophysiology of diabetic kidney disease: impact of SGLT2 inhibitors. Nat Rev Nephrol. 2021 May;17(5):319-334. doi: 10.1038/s41581-021-00393-8. Epub 2021 Feb 5. PMID 33547417